CLINICAL TRIAL: NCT06411366
Title: A Phase I, Open Label, Single Dose Study to Evaluate the Safety and Efficacy of an Injectable Follistatin Plasmid Gene Therapy in Healthy Subjects
Brief Title: Phase I: Safety and Efficacy of an Injectable Follistatin Plasmid Gene Therapy in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Minicircle (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: FST-X7
Record Dates: First submitted 2024-05-08; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Frailty; Aging
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental)
  Interventions: Genetic: Follistatin plasmid

INTERVENTIONS:
Genetic: Follistatin plasmid — Follistatin-344 plasmid

SUMMARY:
This study examines the safety and effects of an injectable plasmid gene therapy. Plasmids are circular pieces of DNA which have been widely studied as a non-permanent & non-heritable method for transferring genes and inducing gene expression. In this study the plasmid is a gene vector which contains the human FST344 gene intended to express and secrete bioidentical human follistatin into serum circulation. Follistatin is a myostatin and activin inhibitor that has demonstrated improved functional outcomes in mouse models of neuromuscular disease.

Participants will undergo dual energy x-ray absorptiometry scans before and after the treatment's administration to compare change from baseline and rates of change in fat vs muscle tissue and bone density. Participants will also undergo metabolic and epigenetic blood panels to observe any changes. Participants will be monitored at the clinic site for a short time period after receiving the therapy and participants will be able to report any adverse events through an online form. Lastly, participants will have blood drawn just prior to, and three months after, the gene therapy's administration in order to assess circulating levels of follistatin. This study is administered at the Global Alliance for Regenerative Medicine clinical research site on the island of Roatan and is sponsored by Minicircle. The main contact for this study is Mac Davis.

ELIGIBILITY:
Inclusion Criteria:

* Openness to morphological change
* Will practice contraception for the duration of trial (if female)

Exclusion Criteria:

* Women who are pregnant, nursing or of childbearing potential who are unwilling or unable to maintain contraceptive therapy for the duration of the study
* Life expectancy < 6 months due to concomitant illness
* Pre-existing joint, ligament, or heart issues
* Systolic blood pressure (supine) ≤90 mmHg;
* Resting heart rate > 100 bpm
* Unwilling or unable to give written informed consent.

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2022-08-18 (Actual); Primary Completion 2023-08-31 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Related Adverse Events as Assessed by CTCAE v4.0 | 3 months
Change from Baseline in Follistatin Serum Concentration at 3 months | 3 months

SECONDARY OUTCOMES:
Change from Baseline in fat-free mass at 3 months via dual x-ray absorptiometry | 3 months
Change from Baseline in fat mass at 3 months via dual x-ray absorptiometry | 3 months
Change in intrinsic and extrinsic epigenetic clock age | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Glenn Terry, MD, Principal Investigator — Principal Investigator
Locations (1):
- Global Alliance for Regenerative Medicine, Roatán, Honduras